CLINICAL TRIAL: NCT02942433
Title: Change Starts at Home: A Cluster Randomized Controlled Trial of a Media and Community Engagement Behavior Change Strategy to Prevent Intimate Partner Violence in Nepal
Brief Title: Intimate Partner Violence Prevention in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Cari Clark, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00091115
Record Dates: First submitted 2016-10-13; First posted 2016-10-24 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radio Program (Experimental): Married couple participants will be asked to interact with a radio program and participate in weekly, sex-separate listening and discussion groups (LDG) that each last for between 75 and 120 minutes over the course of 9 months.
  Interventions: Behavioral: Behavior Change Communication; Behavioral: Community Mobilization; Behavioral: Advocacy
- Control (Other): The control group participants will be exposed to the radio program only, and will not participate in the LDGs, nor will they or their family members participate in the workshops and community activities.
  Interventions: Behavioral: Behavior Change Communication

INTERVENTIONS:
Behavioral: Behavior Change Communication — 9-month weekly episode behavior change radio drama with interactive voice response (IVR)/short message service (SMS) listener engagement
Behavioral: Community Mobilization — Listening and discussions groups, 2 male and 2 female groups per study site meet weekly for 39 weeks and will receive training on gender equity, intimate partner violence (IPV), life skills, community mobilization, non-violent conflict resolution for listening and discussion group (LDG) facilitators to support knowledge and skill set acquisition of LDG members. There will be a joint couple's session every month to foster mutual learning and understanding in addition to community mobilization incentives led by LDGs and encouragement of family members of LGD members to listen to the radio and attend LDG sessions once every 3 months. Participants will also receive awareness raising and street theater to engage families and community members.
  Arms: Radio Program
Behavioral: Advocacy — Training and 6-month follow up of religious/community leaders and religious leaders support community mobilization activity of local listening and discussion group (LGD).
  Arms: Radio Program

SUMMARY:
Introduction: Change Starts at Home (Change) is a multi-component social behavior change communication and community engagement strategy designed to prevent intimate partner violence (IPV), a significant public health issue in Nepal and throughout the world.

Methods and analysis: The study uses a concurrent mixed-methods design. The quantitative aspect of the evaluation is a pair-matched, repeated cross-sectional 2-armed, single-blinded cluster trial (RCT: N=36 clusters, 1440 individuals), comparing a social behavior change communication (SBCC) strategy to radio programming alone for its impact on physical and / or sexual IPV at the end of programming (12 months' post-baseline) and 6-months post the cessation of project activities (24-months post baseline). The qualitative aspects of the design include several longitudinal approaches to understand the impact of the intervention and examine mechanisms of change including in-depth interviews with participants (N=18 couples), and focus group discussions with community leaders (N=3 groups), and family members of participants (N=12 groups). Treatment effects will be estimated with generalized logistic mixed models specified to compare differences in primary outcome from baseline to follow-up, and baseline to 24-months post following intention-to-treat principles.

DETAILED DESCRIPTION:
The Change Starts at Home intervention is a multi-component social behavior change communication (SBCC) strategy designed to shift attitudes, norms and behaviors that underpin the power imbalances between men and women and the perpetration of intimate partner violence (IPV) among couples in Nepal. Recognizing the social ecology of change, the intervention engages actors across multiple rings of influence, such as family members and community leaders, in addition to the primary target audience of married reproductive age women and their husbands. As an SBCC strategy, the intervention approaches intimate partner violence prevention through three key approaches: advocacy, social mobilization and behavior change communication.

Married couple participants will be asked to interact with a radio program and participate in weekly, sex-separate listening and discussion groups (LDG) that each last for between 75 and 120 minutes over the course of 9 months. The same participants will be invited to participate in workshops and community activities such as theater and town hall meetings. Female LDG members will be asked to take a survey three times over the course of 24 months. Family members of LDG members in the treatment condition will be asked to interact with a radio program, and attend up to two focus group discussions (FGD) to understand the environmental facilitators and constraints to the couple exhibiting more gender equitable attitudes and behaviors and changes in family-based norms. Family members will be invited to attend one LDG meeting every 3 months, street theaters and community meetings. Community leaders will be asked to interact with a radio program, to participate in a workshop, to develop a plan of action to promote gender equity and the reduction of violence, to jointly run a community event with an LDG in their area and to attend up to two FGDs. At three separate time points, a randomly selected sample of female community members meeting inclusion criteria will be invited to take a survey.

ELIGIBILITY:
Inclusion Criteria:

Female survey participants

* Of reproductive age (between 18-49 years)
* Husband is at least 18 years of age
* Both the wife and husband reside regularly in the study area
* The wife and husband live together

Family Members

* At least 18 years of age
* A family member of a Listening and Discussion Group member

Community Leaders

* At least 18 years of age
* Considered to be in a position of authority or influence within the study communities per the recommendation of other community stakeholders

Listening and Discussion Group facilitators

* Have a 12th grade standard academic qualification or better
* Be living with his/her spouse
* Have good communication skills
* Have a good reputation in the community based on feedback from local social mobilizers
* Able to commit to 9 months of programming and weekly reporting

Exclusion Criteria:

* Participants must be able to communicate in Nepali
* Must not be have plans to relocate in the coming 2 years
* A physical or cognitive impairment that precludes participation for the duration requested by activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4677 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Change in Prevalence of Physical and/or Sexual Intimate Partner Violence Encounters | Baseline, 24 Month Follow Up
  The number of physical and/or sexual intimate partner violence encounters will be collected via the standard measure for Assessment of Intimate Partner Violence for the Global Program to Prevention Violence Against Women and Girls at baseline, month 12, and month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Cari Clark, Sc.D., M.P.H., Principal Investigator — Emory University

REFERENCES:
- [Derived] Clark CJ, Batayeh B, Shrestha PN, Morrow G, Shrestha B, Ferguson G. Diffusion in social norms change about violence against women: A longitudinal analysis of intervention data from a cluster randomised trial. Glob Public Health. 2021 Oct;16(10):1618-1630. doi: 10.1080/17441692.2020.1828984. Epub 2020 Oct 6. PMID 33021877
- [Derived] Clark CJ, Shrestha B, Ferguson G, Shrestha PN, Calvert C, Gupta J, Batayeh B, Bergenfeld I, Oakes JM. Impact of the Change Starts at Home Trial on Women's experience of intimate partner violence in Nepal. SSM Popul Health. 2019 Dec 13;10:100530. doi: 10.1016/j.ssmph.2019.100530. eCollection 2020 Apr. PMID 31890850
- [Derived] Cardoso LF, Clark CJ, Rivers K, Ferguson G, Shrestha B, Gupta J. Menstrual restriction prevalence and association with intimate partner violence among Nepali women. BMJ Sex Reprod Health. 2018 Sep 28;45(1):38-43. doi: 10.1136/bmjsrh-2017-101908. Online ahead of print. PMID 30266716
- [Derived] Clark CJ, Spencer RA, Shrestha B, Ferguson G, Oakes JM, Gupta J. Evaluating a multicomponent social behaviour change communication strategy to reduce intimate partner violence among married couples: study protocol for a cluster randomized trial in Nepal. BMC Public Health. 2017 Jan 13;17(1):75. doi: 10.1186/s12889-016-3909-9. PMID 28086857